CLINICAL TRIAL: NCT03731546
Title: Effect of Delayed Cord Clamping in Preterm Neonates With Placental Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nehad Nasef, Professor of pediatrics/Neonatology, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS/17.04.15
Record Dates: First submitted 2018-11-03; First posted 2018-11-06 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Preterm Infant; Placental Insufficiency; Placental Transfusion
Keywords: Delayed cord clamping; Preterm Infant; Placental Insufficiency; Intrauterine growth restriction
MeSH Terms: conditions — Premature Birth; Placental Insufficiency; Fetofetal Transfusion; Fetal Growth Retardation | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (No Intervention): Placental insufficiency and ICC : Immediate cord clamping after delivery of the fetus in preterm infants with placental insufficiency
- Group B (Active Comparator): Placental insufficiency and DCC: Cord clamping 60 seconds after delivery of fetus in preterm infants with placental insufficiency
  Interventions: Procedure: Delayed cord clamping
- Group C (Active Comparator): Normal placenta with DCC:Cord clamping 60 seconds after delivery of fetus in preterm infants without placental insufficiency
  Interventions: Procedure: Delayed cord clamping

INTERVENTIONS:
Procedure: Delayed cord clamping — Cord clamping 60 seconds after delivery of fetus in preterm infants
  Arms: Group B; Group C

SUMMARY:
To investigate the effect of delayed cord clamping (DCC) on hematopoietic progenitor cells (HPCs), hematological parameters including haemoglobin concentration and hematocrit value in premature infants (34 weeks gestational age or less) with placental insufficiency.We hypothesized that preterm infants with placental insufficiency underwent DDC could have better hematologic parameters and hematopoietic progenitor cells compared to immediate cord clamping.

DETAILED DESCRIPTION:
• A prospective randomized controlled study will be performed on preterm infants 34 weeks gestational age or less with placental insufficiency, and those without placental insufficiency where DCC will be performed in both groups. A third group of preterm with placental insufficiency and immediate cord clamping will be performed as a control.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates < 34 weeks gestational age

Exclusion Criteria:

* Vaginal bleeding due to placental abruption or tears Multiple pregnancies Suspected major fetal anomalies Suspected chromosomal aberration Maternal drug abuse Hydrops fetalis preterm who needed major resuscitative measures

Ages: 0 Minutes to 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Peripheral venous CD34 at admission | first 24 hours of infants' life
  One milliliter of fetal blood will be taken from peripheral venous blood in the first 30 minutes of life and CD34 will be assessed by flow cytometry.

SECONDARY OUTCOMES:
Admission hemoglobin | first 24 hours of infants' life
  One milliliter of neonatal blood will be taken from peripheral venous blood in the first 24 hours of life.
Hemoglobin at 2 months | 2 months of infants' life
  One milliliter of neonatal blood will be taken from peripheral venous blood at 2 months of life.
Admission platelets | first 24 hours of infants' life
  One milliliter of neonatal blood will be taken from peripheral venous blood in the first 24 hours of life.
Admission WBCs | first 24 hours of infants' life
  One milliliter of neonatal blood will be taken from peripheral venous blood in the first 24
Phototherapy requirements | first 28 days of life
Polycythemia | first 28 days of life
Culture proven sepsis | first 28 days of life
Necrotizing enterocolitis | first 28 days of life
Intraventricular hemorrhage | first 28 days of life
Bronchopulmonary dysplasia | first 70 days of life
Need for nasal CPAP | first 28 days of life
Need for mechanical ventilation | first 28 days of life
Duration of oxygen therapy | first 28 days of life
Need for inotropes | first 28 days of life
Retinopathy of prematurity | first 28 days of life
Need for packed RBCs transfusion | first 28 days of life

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children's Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gokmen Z, Ozkiraz S, Tarcan A, Kozanoglu I, Ozcimen EE, Ozbek N. Effects of delayed umbilical cord clamping on peripheral blood hematopoietic stem cells in premature neonates. J Perinat Med. 2011 May;39(3):323-9. doi: 10.1515/jpm.2011.021. Epub 2011 Mar 11. PMID 21391876
- [Background] Committee on Obstetric Practice, American College of Obstetricians and Gynecologists. Committee Opinion No.543: Timing of umbilical cord clamping after birth. Obstet Gynecol. 2012 Dec;120(6):1522-6. doi: 10.1097/01.AOG.0000423817.47165.48. PMID 23168790
- [Derived] Yunis M, Nour I, Gibreel A, Darwish M, Sarhan M, Shouman B, Nasef N. Effect of delayed cord clamping on stem cell transfusion and hematological parameters in preterm infants with placental insufficiency: a pilot randomized trial. Eur J Pediatr. 2021 Jan;180(1):157-166. doi: 10.1007/s00431-020-03730-4. Epub 2020 Jul 4. PMID 32623628